CLINICAL TRIAL: NCT01914185
Title: The Effectiveness of a Comprehensive School Health Intervention in Improving Healthy Eating and Physical Activity and Preventing Childhood Obesity
Brief Title: Alberta Project Promoting Active Living and Healthy Eating in Schools
Acronym: APPLE Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00003800
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2013-07

CONDITIONS: Childhood Obesity
Keywords: Childhood; Physical activity; Nutrition; Health Promotion
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comparison Schools (No Intervention): Regular health promotion activities
- Comprehensive School Health (CSH) (Experimental): Full time School Health Facilitator present in each school on a day-to-day basis for 3.5 years responsible for facilitating implementation of Comprehensive School Health
  Interventions: Other: Comprehensive School Health (CSH)

INTERVENTIONS:
Other: Comprehensive School Health (CSH) — APPLE Schools uses a CSH approach to health promotion which addresses health through four inter-related pillars 1) positive social and physical environments 2) teaching and learning 3) healthy school policy 4) partnerships and services. A key component of the APPLE Schools intervention was the placement of a full-time School Health Facilitator in each school. Their role was to facilitate the development and implementation of the project, to ensure that it met the schools' unique needs for health promotion, and that it aligned with the core principles of CSH.
  Arms: Comprehensive School Health (CSH)

SUMMARY:
The objectives were to 1) make students eat healthier and be more active; and 2) prevent overweight and obesity. Children will therefore be less likely overweight or obese. Beginning in January 2008, the Alberta Project Promoting active Living and healthy Eating in Schools (APPLE Schools) was implemented in 10 schools throughout the Canadian Province, Alberta. Full-time School Health Facilitators were placed in each of the schools to implement what is know in Canada as Comprehensive School Health (CSH). In the United States, CSH is more commonly referred to as "Coordinated School Health", while the synonymous term "Health Promoting Schools" is often used in Australia and Europe. The project was evaluated annually in the spring from 2008 to 2011 and as of 2009 evaluations included the use of time-stamped pedometers. The comparison group included approximately 150 schools that were randomly selected to reflect the population of Alberta, Canada. Twenty of these randomly selected schools also participated in data collection which involved the use of time-stamped pedometers.

DETAILED DESCRIPTION:
The Alberta Project Promoting active Living and healthy Eating in Schools (APPLE Schools) is a quasi-experimental pre-post trial with a non-equivalent parallel control group. The intervention began in January 2008 and lasted through June 2011 and was implemented school-wide. As out primary interest is to reduce the prevalence of overweight and obesity in schools, the essential comparisons were across grade five students in differing calendar years. At each survey all grade five students were invited to participate. The current design allowed intervention effects to be assessed over time at the school-level. Surveys were administered in the spring of 2008, 2009, 2010, and 2011 in intervention schools. And in the spring of 2008 and 2011 in control schools.

ELIGIBILITY:
Inclusion Criteria:

Intervention Schools:

* school located in a socioeconomically disadvantaged neighbourhood and a demonstrated need for health promotion
* Grade five students with parent consent, who also assented to participate were included in annual evaluations

Control Schools:

* Grade five students with parent consent, who also assented to participate were included in annual evaluations

Exclusion Criteria:

Intervention & Control Schools:

* Schools that did not receive jurisdictional approval to participate
* Grade five students who did not receive parent consent or did not provide their assent were not included in annual evaluations

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8663 (Actual)
Dates: Start 2008-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Overweight and obesity | 24 months
  Students' body weight was measured to the nearest 0.1kg using calibrated digital scales and height was measured to the nearest 0.1cm. BMI was calculated as weight divided by height^2 (kg/m^2). Overweight and obesity were defined using the International Obesity Task Force age and sex specific body mass index (BMI) cut-off points.

SECONDARY OUTCOMES:
physical activity | 24 months
  Children's physical activity was measured using time-stamped pedometers which were worn for 9 consecutive days.
  The Physical Activity Questionnaire for Older Children (PAQ-C) was also used to assess children's physical activity levels
Diet Quality | 24 months
  Students' diet quality was assessed through the use of the Harvard Youth/Adolescent Food Frequency Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Veugelers, PhD, Principal Investigator — University of Alberta
Locations (1):
- Population Health Intervention Research Unit, Edmonton, Alberta, Canada

REFERENCES:
- [Result] Fung C, Kuhle S, Lu C, Purcell M, Schwartz M, Storey K, Veugelers PJ. From "best practice" to "next practice": the effectiveness of school-based health promotion in improving healthy eating and physical activity and preventing childhood obesity. Int J Behav Nutr Phys Act. 2012 Mar 13;9:27. doi: 10.1186/1479-5868-9-27. PMID 22413778
- [Result] Bastian KA, Maximova K, McGavock J, Veugelers P. Does School-Based Health Promotion Affect Physical Activity on Weekends? And, Does It Reach Those Students Most in Need of Health Promotion? PLoS One. 2015 Oct 21;10(10):e0137987. doi: 10.1371/journal.pone.0137987. eCollection 2015. PMID 26488168
- [Result] Vander Ploeg KA, McGavock J, Maximova K, Veugelers PJ. School-based health promotion and physical activity during and after school hours. Pediatrics. 2014 Feb;133(2):e371-8. doi: 10.1542/peds.2013-2383. Epub 2014 Jan 13. PMID 24420806
- [Result] Vander Ploeg KA, Maximova K, McGavock J, Davis W, Veugelers P. Do school-based physical activity interventions increase or reduce inequalities in health? Soc Sci Med. 2014 Jul;112:80-7. doi: 10.1016/j.socscimed.2014.04.032. Epub 2014 Apr 29. PMID 24820223
- [Derived] Dube N, Khan K, Loehr S, Chu Y, Veugelers P. The use of entertainment and communication technologies before sleep could affect sleep and weight status: a population-based study among children. Int J Behav Nutr Phys Act. 2017 Jul 19;14(1):97. doi: 10.1186/s12966-017-0547-2. PMID 28724380
- See also: Related Info — http://appleschools.ca